CLINICAL TRIAL: NCT04340102
Title: Development of a Scalable Intervention to Improve Smoking Cessation in Persons With Serious Mental Illness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Sheppard Pratt Health System (Other); Truth Initiative (Other)
Responsible Party: Principal Investigator, Melanie Bennett, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21CA237468-01A1
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: This project has two phases. Phase 1: Adapt BecomeAnEX, conduct usability testing, and train digital coaches. Phase 2: Implement adapted BecomeAnEx with 60 individuals with a mental health disorder who are hospitalized on the inpatient psychiatric unit at the University of Maryland Medical Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BecomeAnEx (Experimental): Participants will have three individual meetings with a research staff person while they are in the hospital. At these meetings participants will answer questions about their smoking and interest in quitting, learn about BecomeAnEx, and register with the BecomeAnEx program so that they can use it when you leave the hospital. Participants will be given two weeks of nicotine replacement therapy when they leave the hospital. Participants will be asked to use BecomeAnEx as much as they want when they leave the hospital program.
  Interventions: Behavioral: BecomeAnEx

INTERVENTIONS:
Behavioral: BecomeAnEx — This research study is focused on a smoking cessation program called BecomeAnEx. We are studying how to adapt BecomeAnEx for people with a mental health disorder who want to reduce or quit their tobacco smoking. BecomeAnEx includes a website that provides education about smoking and quitting. It also has a text messaging program that delivers personalized information. Persons in the program have access to real-time digital coaching with a remote coach who has experience helping people quit smoking. In addition, the program has an on-line community of current and former smokers that can provide support and encouragement.

SUMMARY:
All patients with serious mental illness are abstinent while in the hospital for a psychiatric admission yet almost all return to smoking after discharge. The investigators propose to adapt a digital intervention both to the needs of SMI smokers and to being introduced in the inpatient psychiatric setting through a collaboration between experts in SMI and the Truth Initiative, a pre-eminent tobacco control organization. The investigators believe this will bridge the inpatient to outpatient gap in cessation services and will help people remain abstinent following hospital discharge.

DETAILED DESCRIPTION:
Persons with serious mental illness (SMI, schizophrenia, bipolar disorder, recurrent depression) are a socioeconomically disadvantaged group and die on average 10-15 years earlier than those in the general population, many from cancer. The prevalence of smoking in persons with SMI is approximately 3 times that in the general population; smoking is the is the strongest risk factor for elevated mortality in this population. Psychiatric inpatient admissions are common in SMI and the hospital is an optimal place to provide smoking cessation services. All patients are abstinent while in the hospital. The key challenge is how to continue to engage these patients in cessation services to support continued abstinence. While most receive refer to telephone quitline at discharge, quitlines are not as effective with SMI smokers and almost all return to smoking. Introducing hospitalized SMI patients to cessation services that can be easily accessed when they leave the hospital offers the best chance of converting initial abstinence into sustained abstinence post-discharge. A digital intervention that incorporates web-delivered evidence-based smoking cessation practices, digital coaching, and mobile text messaging is a scalable and sustainable way to bridge the inpatient to outpatient gap in cessation services. Currently there is no digital cessation program that addresses the needs of SMI smokers. The investigators propose to adapt a digital intervention both to the needs of SMI smokers and to being introduced in the inpatient psychiatric setting through a collaboration between experts in SMI and the Truth Initiative, a pre-eminent tobacco control organization. The investigators will build upon a well-established, evidence-based, cessation website, BecomeAnEX.org (EX), that offers individualized quit plans, an active social community, text and email messaging support, and digital coaching. Integrating input from different stakeholders, the investigators will develop adaptations so that EX components and language are in line with principles of mental health recovery and will successfully engage SMI smokers with digital coaching that will support use of other EX services. The investigators will develop automated and integrated procedures for identifying hospitalized SMI smokers and registering them with EX. The investigators will then examine the feasibility and acceptability of the adapted intervention to engage and retain 60 smokers with SMI after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Diagnosis of serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder, or major depression)
* Current smoker [prior to admission, smoked at least one cigarette or small cigar per day in the past month (unless restricted, e.g. due to ER/hospital visit) and smoked at least 100 cigarettes lifetime]
* Interested in remaining quit after hospital discharge or quitting within the following 30 days
* Expected Internet use at least several times a week post-discharge and ownership of mobile device with text messaging plan post-discharge
* Sufficiently stable and cooperative to engage in the intervention, operationalized as not on a nursing observation level that indicates high acuity/safety concerns and has participated in a majority of hospital unit activities as documented in the chart during the hospital stay so far

Exclusion Criteria:

* Intellectual disability (DSM5 317, 318), traumatic brain injury, or deafness.
* Homeless prior to admission or anticipated to be homeless at discharge.
* Discharge to a residential setting where smoking is prohibited.
* Medical condition for which the use of nicotine replacement therapy (NRT) is contraindicated including pregnant, planning to become pregnant, or breastfeeding; within 4 weeks post myocardial infarction; severe arrhythmia, severe angina pectoris; peptic ulcer; severe renal failure; poorly controlled insulin-dependent diabetes; severely uncontrolled hypertension; peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 2 months
  Rate of recruitment
Feasibility of registration | 2 months
  Time to register with the web based intervention
Acceptability | 2 months
  Satisfaction with the web based intervention using the Client Satisfaction Questionnaire
Acceptability | 2 months
  Satisfaction with the web based intervention using the Services Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No